CLINICAL TRIAL: NCT02511600
Title: A Randomized Phase III Trial to Compare the Progel Sealant to Standard of Care (SOC) for Patients Undergoing Decortication for Mesothelioma or Other Pathologies
Brief Title: Comparison of Progel Sealant to Standard of Care (SOC) for Patients Undergoing Decortication
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bard Incorporated (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-0958; NCI-2015-01511 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-07-28; First posted 2015-07-30 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Lung Diseases; Mesothelioma
Keywords: Lung Diseases; Mesothelioma; Pleurectomy decortication; Progel; Talcum powder; Pain questionnaires; Surveys; Intraoperative air leaks; IAL
MeSH Terms: conditions — Lung Diseases; Mesothelioma | interventions — Talc; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Progel Sealant (Experimental): After pleurectomy decortication, Progel® sealant added to the surface of the lung prior to closure of the chest. Participants complete pain scale 3 times each day while in the hospital.
  Interventions: Other: Progel Sealant; Behavioral: Pain Questionnaire
- Standard of Care (Active Comparator): After pleurectomy decortication, talcum powder added to the surface of the lung prior to closure of the chest. Participants complete pain scale 3 times each day while in the hospital.
  Interventions: Other: Talcum Powder; Behavioral: Pain Questionnaire

INTERVENTIONS:
Other: Progel Sealant — After pleurectomy decortication, Progel® sealant added to the surface of the lung prior to closure of the chest.
  Arms: Progel Sealant
Other: Talcum Powder — After pleurectomy decortication, talcum powder added to the surface of the lung prior to closure of the chest.
  Arms: Standard of Care
Behavioral: Pain Questionnaire — Participants complete pain scale 3 times each day while in the hospital. Pain is rated on a pain scale of 0 - 10.
  Other Names: Survey

SUMMARY:
The goal of this clinical research study is to compare Progel® (a type of surgical sealant that is made from human blood products) to the standard of care (talcum powder) to learn if one method is better than the other for preventing air leaks in patients having a pleurectomy decortication.

DETAILED DESCRIPTION:
If participant agrees to take part in this study, they will have their pleurectomy decortication as planned. Participant will sign a separate consent for this procedure that explains the risks.

At the time of participant's surgery, sutures and staples are used to help correct air leaks, which is standard.

Then, participant will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups. This is done because no one knows if one study group is better, the same, or worse than the other group:

* One group will have Progel® added to the surface of the lung before closing the chest.
* The other group will have talcum powder added to the surface of the lung before closing the chest.

Participant will have an equal chance of being in either group.

During the surgery, air leaks will be checked electronically and that information will be recorded.

After surgery, participant will be asked to rate their pain on a pain scale of 0-10. Participant will be asked to complete this pain scale 3 times each day while they are in the hospital.

Length of Study Participation:

After participant's surgery and their air leak is resolved, their participation in this study will be over.

This is an investigational study. The Progel® surgical sealant is FDA approved for the control of air leaks during lung surgery. It is investigational to compare the surgical sealant with the standard-of-care (talcum powder) to learn if it can reduce the number of days in the hospital after surgery.

Up to 48 participants will enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with mesothelioma or other pathologies undergoing a pleurectomy decortication at MD Anderson Cancer Center
2. Adequate preoperative renal function documented by serum creatinine of < 1.5 mg/dl or calculated creatinine clearance > 50 ml/min

Exclusion Criteria:

1. Patients unable to consent for the procedure
2. Patients with a history of allergy to human proteins
3. Patients who may have insufficient renal capacity for clearance of Progel® polyethylene glycol load

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Time to Resolve Air Lung Leak After Pleurectomy Decortication | Participants followed for the duration of hospital stay, at least 5 days.
  Primary outcome is T = time to resolve an air leak in the lungs, allowing the possibility that an air leak may not develop, represented by T=0.

CONTACTS AND LOCATIONS:
Overall Officials: Reza J. Mehran, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org